CLINICAL TRIAL: NCT00259623
Title: Efficacy at 3 Months on Permanent Atrial Fibrillation in Patients Candidates to Cardiac Surgical Treatment by Epicardial, or Possibly Endocardial, Radiofrequency Ablation
Brief Title: Cardiac Surgical Treatment by Radiofrequency Ablation on Valvular Patients: Efficacy at 3 Months
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Roques, University Hospital Toulouse
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0406902; AOL
Record Dates: First submitted 2005-11-25; First posted 2005-11-29 (Estimated); Last update posted 2009-07-17 (Estimated); Status verified 2009-07

CONDITIONS: Atrial Fibrillation
Keywords: Cardiac surgery; Radiofrequency ablation; Atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Radiofrequency ablation

SUMMARY:
The objective of the study is to evaluate the efficacy of the epicardial or endocardial radiofrequency ablation in the treatment of atrial fibrillation.

It is a multicentric, prospective, randomized, parallel, comparative, double blind study. The study principal objective is to evaluate the absence of atrial fibrillation after 3 months. The secondary objectives consist in the evaluation of the maintenance of the sinusal heart rate at one year and of the quality of life improvement

DETAILED DESCRIPTION:
Principal objective:

To evaluate the efficacy at 3 months of combined ablation technique in the treatment of chronic atrial fibrillation during cardiac surgery in order to obtain a sinusal heart rate.

A sequential statistical analysis of the results will be performed every 10 patients.

In case of validation of the principal objective by a sequential method i.e. proving the superiority of the treatment by ablation, ,the study would then be opened and pursued by using the ablation technique for all subsequent patients in order to validate the secondary study objectives

Secondary objectives:

* To evaluate the quality of life of the patients at one year and the absence of atrial fibrillation relapse.
* 6 and 12 months clinical follow-up
* To evaluate the left atrial function at 6 months by trans-oesophagus echocardiography

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with no age limit, presenting a chronic atrial fibrillation and planned to undergo a surgical intervention on mitral valve (valve replacement or plasty) associated or not with myocardial revascularization or replacement/plasty of another valve (aortic, tricuspid)
* The chronic atrial fibrillation is defined as a continuous atrial fibrillation more than 1 month before the surgery despite all anti-arrhythmia treatments including cardioversion ; the atrial fibrillation can be associated to another rhythm trouble except the severe ventricular rhythm troubles.
* The indication for surgery is performed using the clinical evaluation : NYHA >2 and the usual echocardiography criteria (mitral regurgitation > grade 3, mitral gradient >10 mm Hg or valve surface < 1,5 cm2)
* Patients with a vital prognosis not compromised by comorbidity in the next 2 years and with a mental state enabling to give informed consent
* Patients agreeing to take part in the study and having signed the informed consent form.

For the part of the study pursued in open independent to the actual protocol, patients having signed the modified informed consent with approval of the new study procedure not yet published.

Exclusion Criteria:

* Paroxystic atrial fibrillation or atrial fibrillation for less than 1 month
* Atrial fibrillation never treated by cardioversion or pharmacology before surgery.
* Contra-indication to surgery, i.e. severe respiratory failures, multivisceral deficiencies (renal, cardiac or hepatic), rapidly evolutive or metastatic cancers, malignant hemopathies not stabilized by chemotherapy
* Contra-indication to the following arrhythmia treatments: class III (amiodarone) associated to contra-indication to class II (beta blockers) or to class Ic (flecainide, propafenone, cibenzoline).
* Severe decompensated heart failure.
* Uncontrolled, repetitive, severe documented ventricular arrhythmia (ventricular tachycardia, ventricular fibrillation episodes)
* Contra indication to epicardic ablation procedure (pericardic adhesions, intra-atrial thrombus) In these cases the ablation could be only an endocardic ablation but it does not necessarily exclude the patient.
* Ventricular "ejection fraction " < 40%
* Impossibility to follow the pre-inclusion phases i.e. emergency surgery for mitral break or evolutive endocarditis.
* Patients with disabled mental status
* Patient participating in another clinical study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2005-12; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
- absence of atrial fibrillation at 3 months.
The patients presenting a spontaneous sinus rhythm heart rate or who need a permanent pace maker at 3 months will be considered as SUCCESSFUL.
The patients presenting at 3 months either an atrial fibrillation or a left flutter despite an adapted anti-arrythmia treatment and one electric cardioversion,and the patients who died before the 3 months evaluation will be considered as FAILURES

CONTACTS AND LOCATIONS:
Overall Officials: Gérard FOURNIAL, MD, Principal Investigator — University Hospital, Toulouse, France
Locations (5):
- France (5):
  - Service de Chirurgie Cardio-Vasculaire - Hôpital Côte de Nacre, Caen, CAEN
  - Service de Chirurgie Cardio-Vasculaire - Hôpital Gabriel Montpied, Clermont-Ferrand, Clermont-ferrand
  - Service de Chirurgie Cardio-vasculaire - CHU Dupuytren, Limoges, Limoges
  - Service de Chirurgie Cardio Vasculaire - CHU RANGUEIL, Toulouse, Toulouse
  - Service de Chirurgie Cardio Vasculaire - Clinique Pasteur, Toulouse, Toulouse

REFERENCES:
- [Background] Benussi S, Nascimbene S, Agricola E, Calori G, Calvi S, Caldarola A, Oppizzi M, Casati V, Pappone C, Alfieri O. Surgical ablation of atrial fibrillation using the epicardial radiofrequency approach: mid-term results and risk analysis. Ann Thorac Surg. 2002 Oct;74(4):1050-6; discussion 1057. doi: 10.1016/s0003-4975(02)03850-x. PMID 12400744
- [Result] Raman JS, Ishikawa S, Power JM. Epicardial radiofrequency ablation of both atria in the treatment of atrial fibrillation: experience in patients. Ann Thorac Surg. 2002 Nov;74(5):1506-9. doi: 10.1016/s0003-4975(02)03945-0. PMID 12440600